CLINICAL TRIAL: NCT03966469
Title: Informed Consent for Pelvic Reconstruction: Does Having a Support Person Matter
Brief Title: What is the Impact of the Presence of a Support Person on Informed Consent
Status: Completed | Type: Observational
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Sappenfield, Principle Investigator, Hartford Hospital
Other Study IDs: HHC-2018-0251
Record Dates: First submitted 2019-05-17; First posted 2019-05-29 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Surgery; Knowledge, Attitudes, Practice; Prolapse, Vaginal; Urinary Incontinence
Keywords: informed consent; support person
MeSH Terms: conditions — Behavior; Uterine Prolapse; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Support Person Present: Participants who bring a support person with them to their preoperative appointment.
  Interventions: Other: Preoperative support person present
- Patient Present Only: Participants who present by themselves to their preoperative appointment.
  Interventions: Other: Patient Present Only

INTERVENTIONS:
Other: Preoperative support person present — Participants who bring a support person to their preoperative appointment.
  Groups: Support Person Present
Other: Patient Present Only — Patient presents to their preoperative appointment without a support person.
  Groups: Patient Present Only

SUMMARY:
In practice, the Investigators recommend that patients bring a family member or close friend to their pre-operative appointment to help with patient anxiety, comprehension, and informed decision-making. However, there is limited literature to support this recommendation. The investigators are exploring if having a support person present during this consent process impacts anxiety, satisfaction, knowledge, and preparedness for surgery.

DETAILED DESCRIPTION:
Introduction:

In practice, the investigators recommend that patients bring a family member or close friend to their pre-operative appointment to help with patient anxiety, comprehension, and informed decision-making. However, there is limited literature to support this recommendation. The investigators hypothesize that having a family member or close friend present will decrease patient anxiety and improve patient satisfaction and recall regarding the risks/benefits/ alternatives of surgery.

Study Objectives The primary objective is to assess the impact of having a support person present during the patient's preoperative visit on patient anxiety regarding informed consent for surgery. The secondary objective is to assess the impact of a support person on patient satisfaction, self-assessment of understanding, knowledge, time spent with patient, and pre- and post-operative phone calls.

Hypotheses HO: For women with a support person present during their preoperative visit, there is no difference in the patient-reported anxiety regarding informed consent for surgery compared with women without a support person present.

HA: For women with a support person present during their preoperative visit, there is a difference in the patient-reported anxiety regarding informed consent for surgery compared with women without a support person present.

Research Questions

The research questions to be answered as a part of this study are:

Does having a support person present at the pre-operative visit affect anxiety, satisfaction, preparedness and knowledge regarding their surgery? Does having a support person present impact utilization of clinic resources including preoperative phone calls, and postoperative phone calls?

Study Design and Methods This study will be a prospective cohort study. All women scheduled to undergo vaginal pelvic reconstructive surgery will be recruited from the Urogynecology clinics of the Hartford Hospital Medical Group at the time of their pre-operative appointment. Patients who qualify for inclusion and consent to participate will be enrolled in the study.

Participants will be assigned to one of two arms:

the "support person present" arm, or the "patient present only" arm.

Participants will answer questionnaires prior to their appointment with the physician, after the appointment, 2-3 days prior to surgery via telephone, and at their postoperative appointment.

Risks/Benefits to Patients This is a minimal-risk study. The only research element, and therefore introduction of potential risk(s) beyond standard-of-care treatment, comprises administration of several surveys and data collection.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a 23-hr observation or inpatient surgery for pelvic organ prolapse
* Able to understand English
* Able/willing to sign the informed consent document

Exclusion Criteria:

* Surgery canceled
* Inability to provide consent
* Resident of a long-term care facility or utilization of a home health service
* Scheduled for outpatient surgery
* non-English speaking
* unable/unwilling to sign informed consent document

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women planning to undergo pelvic organ prolapse surgery with our Urogynecology team.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety | Immediately prior to the preoperative visit with the physician and immediately after the preoperative appointment.
  We will measure anxiety with the Spielberger State-Trait Anxiety Inventory (STAI-6) questionnaire. Score ranges from 20 to 80 with higher values indicating higher anxiety.

SECONDARY OUTCOMES:
Patient satisfaction immediately after the preoperative appointment: the Satisfaction with Decision Scale for Pelvic Floor Disorders (SDS-PFD) questionnaire | Patient satisfaction measured immediately after the preoperative appointment prior to leaving the clinic.
  We will measure satisfaction with the SDS-PFD questionnaire. The SDS-PFD is composed of 6 individual items graded from 1 to 5, with higher scores indicating higher satisfaction.
Patient satisfaction prior to surgery: the Satisfaction with Decision Scale for Pelvic Floor Disorders (SDS-PFD) questionnaire | Patient satisfaction measured via telephone 2-3 days prior to surgery.
  We will measure satisfaction with the SDS-PFD questionnaire. The SDS-PFD is composed of 6 individual items graded from 1 to 5, with higher scores indicating higher satisfaction.
Preparedness at the preoperative appointment | Immediately after the preoperative appointment, the preparedness questionnaire will be provided
  We will measure preparedness with the preoperative preparedness questionnaire. This is an 11 item questionnaire graded from 1 to 6, with lower scores indicating higher preparedness.
Preparedness 2-3 days prior to surgery | 2-3 days prior to scheduled surgery, participants will be called and a preparedness questionnaire asked.
  We will measure preparedness with the preoperative preparedness questionnaire. This is an 11 item questionnaire graded from 1 to 6, with lower scores indicating higher preparedness.
Knowledge after the preoperative appointment | Immediately after the the preoperative appointment involving informed consent.
  We will measure knowledge with a knowledge questionnaire. This is a 14 item questionnaire graded in a yes/no format with lower scores indicating lower knowledge.
Knowledge 2-3 days prior to surgery | 2-3 days prior to surgery, participants will receive a phone call where we will ask questions regarding knowledge (complete the knowledge questionnaire)
  We will measure knowledge with a knowledge questionnaire. This is a 14 item questionnaire graded in a yes/no format with lower scores indicating lower knowledge.
Phone calls. | From time of enrollment up to the participants 3-5 week postoperative appointment.
  We will monitor the incidence of phone calls prior to and after surgery by chart review.
Postoperative satisfaction: questionnaire | At the 3-5 week postoperative appointment.
  We will measure postoperative satisfaction with a postoperative satisfaction questionnaire. This is a 7 item questionnaire with lower scores indicating higher satisfaction/preparedness.
Impression of improvement at postoperative appointment | At the 3-5 week postoperative appointment, patients will be provided the PGI-I questionnaire
  We will measure impression of improvement with a Patient Global Impression of Improvement Questionnaire. This is a 1 item questionnaire graded from 1 to 7, with lower scores indicating greater postoperative improvement condition.
Anxiety prior to surgery | 2-3 days prior to surgery
  We will call participant several days prior to surgery and ask Spielberger State-Trait Anxiety Inventory (STAI-6) over the phone. Score ranges from 20 to 80 with higher values indicating higher anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not available to other researchers.

REFERENCES:
- [Derived] Sappenfield EC, O'Sullivan DM, Steinberg AC. The Value of a Support Person During the Surgical Consent Process: A Prospective Cohort Study. Female Pelvic Med Reconstr Surg. 2022 Jan 1;28(1):27-32. doi: 10.1097/SPV.0000000000001059. PMID 34978544

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03966469/Prot_SAP_000.pdf